CLINICAL TRIAL: NCT07078474
Title: Comparison of Different Methods of Hyaluronic Acid Application on Skin Parameters
Brief Title: Comparison of Skin Condition After Hyaluronic Acid Application on Dry vs. Moist Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2181-198-03-04-25-0064
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Skin Hydration; Hyaluronic Acid
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Skin Application (Experimental): Participants in this group applied hyaluronic acid topically to clean, dry skin. The aim was to evaluate hydration and skin parameter changes following this method of application.
  Interventions: Other: Topical Hyaluronic Acid
- Moist Skin Application (Experimental): Participants in this group applied hyaluronic acid topically to pre-moistened skin. The goal was to assess whether applying the product to damp skin enhances its hydrating effect.
  Interventions: Other: Topical Hyaluronic Acid

INTERVENTIONS:
Other: Topical Hyaluronic Acid — Hyaluronic acid was applied topically to the facial skin of healthy participants once daily for a period of 3 weeks. Two application methods were used: on dry skin and on pre-moistened skin. Skin measurements were performed at baseline and after each week of intervention (Week 1, Week 2, and Week 3) to assess hydration and other skin parameters.

SUMMARY:
This study aims to compare the effects of two different methods of applying hyaluronic acid (HA) on skin parameters in healthy individuals. HA is a widely used ingredient in skincare products due to its hydrating properties. However, it is unclear whether applying HA to dry or pre-moistened skin provides better results in terms of skin hydration and texture.

In this non-invasive, interventional trial, 23 healthy volunteers aged 18 to 50 will be randomly assigned to two groups. One group will apply HA to dry skin, while the other will apply HA to moistened skin. Skin parameters will be measured before and after the intervention to assess hydration, transepidermal water loss, and overall skin condition.

The aim is to determine the optimal method of HA application that maximizes its effectiveness in improving skin quality. Participants may benefit from improved skin hydration and increased awareness of the best application method for their skin type. No significant risks are expected from participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18 to 50 years
* Willingness to apply the product daily for 3 weeks
* Ability to attend all scheduled skin assessments (baseline + weekly)
* Provided written informed consent

Exclusion Criteria:

* Known allergy or sensitivity to hyaluronic acid or any component of the product
* Active skin diseases or dermatological conditions in the facial area
* Use of systemic or topical corticosteroids or retinoids within 4 weeks prior to study
* Pregnancy or breastfeeding
* Participation in another clinical trial within the past 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change in skin hydration level | Baseline, Week 1, Week 2, Week 3
  Skin hydration will be measured at four time points using a corneometer or comparable non-invasive skin analysis device. Measurements will be taken before the intervention (baseline) and at the end of each week to assess cumulative and comparative effects of hyaluronic acid application.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Split School of Medicine, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: No